CLINICAL TRIAL: NCT01297400
Title: Phase 2 Pilot Study of the Safety and Efficacy of Topical MW-III in Thermal Burns
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Skingenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MW-III-BURN-2-001
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Burns
Keywords: Burns, Partial Thickness Burns
MeSH Terms: conditions — Burns | interventions — Drugs, Investigational; Silver Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Drug, MW-III (Experimental): Investigational Drug, MW-III
  Interventions: Drug: Investigational Drug, MW-III
- Standard of care (Active Comparator): Silvadene® Cream 1% [Silver Sulfadiazine]
  Interventions: Drug: Silvadene® Cream 1% [Silver Sulfadiazine]

INTERVENTIONS:
Drug: Investigational Drug, MW-III — Topical application, twice a day
  Arms: Investigational Drug, MW-III
Drug: Silvadene® Cream 1% [Silver Sulfadiazine] — Topical application, twice a day
  Arms: Standard of care

SUMMARY:
To compare MW-III to Silvadene® Cream 1% (Silver Sulfadiazine) with respect to "time to healing" (≥95% re-epithelialization) of a partial thickness target thermal burn.

DETAILED DESCRIPTION:
This phase 2 pilot study will assess the safety and efficacy of topical MW-III on thermal burns.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years of age or older on the day of signing the informed consent.
2. Thermal Burns not exceeding a total body surface area (TBSA) OF 25%, with at least one partial thickness burn of 0.5% TBSA or greater. If full thickness burn(s) are present at screening, the total full thickness burn area shall not exceed 10% TBSA. Note: TBSA excludes areas of superficial (first degree) burns.
3. Able and willing to give informed consent and comply with study procedures.

Exclusion Criteria:

1. Any burn that at screening is:

   1. infected.
   2. circumferential or deemed, in the judgment of the investigator, at high risk for developing compartment syndrome.
   3. partial thickness that is likely, in the judgment of the Investigator, to require grafting within 72 hours, or other non-protocol intervention.
2. Severe inhalation injury or other significant non-burn trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to healing (≥95% re-epithelialization) of the partial thickness target burn. | 28 days Treatment Period
  Time to healing (≥95% re-epithelialization) of the partial thickness target burn.

SECONDARY OUTCOMES:
Proportion of subjects with partial thickness burns that are healed at each scheduled study assessment. | 28 days Treatment Period
  Proportion of subjects with partial thickness burns that are healed at each scheduled study assessment.
Proportion of subjects with partial thickness burns determined by PI to require skin grafting of burn wound by Day 28. | 28 days Treatment Period
  Proportion of subjects with partial thickness burns determined by PI to require skin grafting of burn wound by Day 28.
Scar scores (POSAS) of the partial thickness target burn and all other partial thickness burns at Day 28. | 28 days Treatment Period
  Scar scores (POSAS) of the partial thickness target burn and all other partial thickness burns at Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Foster, Principal Investigator — Valleywise Health Medical Center
Locations (6):
- United States (4):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - University of CA Davis Medical Center, Sacramento, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Iowa Health Care, Iowa City, Iowa
- Mexico (2):
  - Proactive CR Mexico SA de CV, Irapuato
  - SMIQ S de R. L de CV, Querétaro City

IPD SHARING:
Plan to Share IPD: No